CLINICAL TRIAL: NCT07241377
Title: A Randomized, Double-blind Placebo-controlled Study in Healthy Subjects to Compare the Bioavailability of EPA + DHA From Two Microalgal Sources in Natural Triglyceride Form to One Fish Source in Re-esterified Triglyceride Form (GOBO 2 Study)
Brief Title: A Study in Healthy Adults to Compare the Bioavailability of EPA + DHA From Two Microalgal Sources to One Fish Source and Placebo
Acronym: GOBO 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: DSM-Firmenich AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024-20-08-GOBO2
Record Dates: First submitted 2025-09-22; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Absorption of Omega-3; Omega-3 Supplementation; Healthy Participants
Keywords: GOBO 2; Omega-3; Fish oil; microalgal oil
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- life'sTM Omega O1035DS nTG (Experimental): life'sTM Omega O1035DS is a nTG derived from microalgae with minimum 365 mg DHA, minimum 100 mg EPA, and minimum 520 mg/g DHA + EPA. All Omega-3 oils will be diluted with high oleic sunflower oil for a total (EPA + DHA) content of 300 mg/capsule. Each subject will consume three capsules for a total intake of 900 mg (EPA+DHA)/day for 6 weeks.
  Interventions: Dietary Supplement: life'sTM omega O1035DS nTG
- life'sTM Omega O3020DS nTG (Experimental): life'sTM Omega O3020DS is a nTG derived from microalgae with minimum 210 mg DHA, minimum 300 mg EPA, and minimum 510 mg/g DHA + EPA. All Omega-3 oils will be diluted with high oleic sunflower oil for a total (EPA + DHA) content of 300 mg/capsule. Each subject will consume three capsules for a total intake of 900 mg (EPA+DHA)/day for 6 weeks.
  Interventions: Dietary Supplement: life'sTM omega O3020DS nTG
- MEG-3TM 3223 rTG (Active Comparator): The fish oil will be MEG-3TM 3223 rTG with minimum 230 mg DHA, minimum 320 mg EPA, and minimum 640 mg/g Omega-3. All Omega-3 oils will be diluted with high oleic sunflower oil for a total (EPA + DHA) content of 300 mg/capsule. Each subject will consume three capsules for a total intake of 900 mg (EPA+DHA)/day for 6 weeks.
  Interventions: Dietary Supplement: MEG-3 3323rTG
- Placebo (Placebo Comparator): The placebo capsules will be a mixture of corn and soybean oils. 515 mg corn oil and 515 mg soybean oil. Each subject will consume three capsules for a day for 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: life'sTM omega O1035DS nTG — All Omega-3 oils will be diluted with high oleic sunflower oil for a total (EPA + DHA) content of 300 mg/capsule. Each subject will consume three capsules for a total intake of 900 mg (EPA+DHA)/day for 6 weeks.
  Other Names: Microalgal oil
  Arms: life'sTM Omega O1035DS nTG
Dietary Supplement: life'sTM omega O3020DS nTG — All Omega-3 oils will be diluted with high oleic sunflower oil for a total (EPA + DHA) content of 300 mg/capsule. Each subject will consume three capsules for a total intake of 900 mg (EPA+DHA)/day.
  Other Names: Microalgal oil
  Arms: life'sTM Omega O3020DS nTG
Dietary Supplement: MEG-3 3323rTG — All Omega-3 oils will be diluted with high oleic sunflower oil for a total (EPA + DHA) content of 300 mg/capsule. Each subject will consume three capsules for a total intake of 900 mg (EPA+DHA)/day.
  Other Names: Fish oil
  Arms: MEG-3TM 3223 rTG
Other: Placebo — The placebo capsules will be a mixture of corn and soybean oils. 515 mg corn oil and 515 mg soybean oil. Each subject will consume three capsules a day.
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, parallel, placebo-controlled study in healthy adults to compare the absorption of two microalgal formulations, to a fish oil and a placebo. Participant will take their assigned study product for 6 weeks and attend the clinic for 4 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any trial related assessments are performed.
2. Healthy adult females ages 18-64 who are neither pregnant nor breastfeeding or healthy adult males ages 18-64 at the time of consent.

   a. Female participants of child-bearing potential (females who are post-menopausal, i.e., when there has been no menstruation for a minimum of 12 months prior to screening, are considered not to be of child-bearing potential), who are not surgically sterilized, must have a negative pregnancy test at screening and be willing to practice one of the following appropriate contraceptive methods until the last visit: i. Sexual abstinence. ii. Oral contraceptives. iii. Trans dermal patches or depot injection of a progestogen drug (starting at least 4 weeks prior to product administration).

   iv. Intrauterine device (IUD), intrauterine system (IUS), subdermal implant, or vaginal ring (placed at least 4 weeks prior to product administration).

   v. Contraceptives must be effective before the randomization visit.
3. Participant's body mass index (BMI) must be between 18 and 30 kg/m2 (inclusive) and participant must weigh a minimum of 50 kg (110 lbs).
4. Intakes of EPA+DHA of <200 mg per day based on the FFQ
5. Agree not to change current diet and exercise frequency or intensity during entire study period

Exclusion Criteria:

1. Participant has any health conditions that would prevent from fulfilling the study requirements, put the participant at risk or would confound the interpretation of the study results as judged by the Investigator based on medical history and routine laboratory test results.
2. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
3. Has a clinically significant abnormal finding on the medical assessment, medical history, vital signs or clinical laboratory results at screening.
4. History or presence of allergic or adverse response to omega-3-acid ethyl esters or triglycerides (EPA or DHA), or related drugs, or sensitivity or allergy to fish or shellfish, or soybean or corn.
5. History of coagulation disorder or current anticoagulation therapy.
6. Has been on a significantly abnormal* diet, as deemed by the investigator, during the 4 weeks preceding the first dose of study medication. *an abnormal diet will be considered if the participant has elected to change to a more or less restricted diet of any description (e.g., change to or from a vegetarian, vegan, gluten-free, lactose-free, etc.) or significantly increases or decreases their daily caloric intake.
7. Has participated in another clinical trial (randomised participants only) within 30 days prior to the first dose of study medication.
8. Has used prescription medication (excluding oral contraceptive and hormonal replacement therapy) within 4 weeks of screening or OTC medication within 7 days before the first dose that may affect omega-3 absorption or any study outcomes. This may include but is not limited to: high-dose NSAIDs, bile acid sequestrants, statins, GLP-1 receptor agonists, anticoagulants and anti-inflammatory drugs. Occasional ibuprofen, paracetamol and low-dose aspirin use is permitted.
9. Regular use* of omega-3 supplements and/or regular fatty fish consumption within 2 months. *Regular use is defined as more than once per week of either fish oil, krill oil, microalgal oil supplements, or fatty fish.
10. Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
11. History of substance abuse or treatment (including more than 14 alcoholic drinks per week) within the past 2 years based on the judgement of the investigator.
12. Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).
13. Has increased bleeding from existing pathological conditions or anticipates surgery (including dental) prior to, throughout, or within 1 week after study participation.
14. Has had a transient ischemic attack (TIA) or stroke or is at high risk for recurrent ischemic events

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The change in plasma phospholipids EPA+DHA µg/ml levels from baseline to week 6 between MEG-3 3223, O1035DS nTG and O3020DS nTG and placebo | Baseline to week 6
  The change in plasma phospholipids EPA+DHA µg/ml levels from baseline to week 6 between MEG-3 3223, O1035DS nTG and O3020DS nTG and placebo as determined by Gas Chromatography (GC).

SECONDARY OUTCOMES:
To compare the bioavailability of Omega-3 fatty acids after the supplementation of O1035DS nTG, O3020DS nTG, MEG-3 3223rTG to placebo by comparing the changes from baseline in the sum level of plasma phospholipids at 2, 4 and 6 weeks of supplementation. | Baseline, week 2, week 4, week 6
  The change in plasma phospholipids EPA+DHA µg/ml levels from baseline to week 2, 4, and 6 between MEG-3 3223 rTG, O1035DS nTG, O3020DS nTG and placebo as determined by Gas Chromatography (GC).
To compare the bioavailability of Omega-3 fatty acids (EPA+DHA) from MEG-3 3223, O1035DS nTG, O3020DS nTG to placebo by comparing the change from baseline in the Omega-3 Index at the end of 6 weeks supplementation. | Baseline to week 6
  The change in the Omega-3 Index from baseline to week 6 between MEG-3 3223, O1035DS nTG, O3020DS nTG and placebo as determined by Gas Chromatography (GC).
To assess the bioavailability of Omega-3 fatty acids after the supplementation of MEG-3 3223, O1035DS nTG, O3020DS nTG and placebo by comparing the changes in the sum level of plasma phospholipids from baseline at 2 and 4 weeks of supplementation. | Baseline, week 2, week 4
  The change in plasma phospholipids EPA+DHA µg/ml levels from baseline to week 2 and 4 after supplementation of MEG-3 3223, O1035DS nTG, O3020DS nTG and placebo as determined by Gas Chromatography (GC).
To compare changes from baseline in lipoprotein levels (total cholesterol, HDL- and LDL-cholesterol and triglyceride levels) after supplementation of MEG-3 3223, O1035DS nTG, O3020DS nTG and placebo at the end of a 6-week study. | Baseline, week 6
  The change in total cholesterol, HDL- and LDL-cholesterol and triglyceride levels from baseline to week 6 between MEG-3 3223, O1035DS nTG, O3020DS nTG and placebo as determined by a clinical analyser.

OTHER OUTCOMES:
Additional 1: Change from baseline in plasma phospholipid EPA at weeks 2, 4 and 6 across the groups adjusted for intake level | Baseline, week 2, week 4, week 6
  Change from baseline in plasma phospholipid EPA at weeks 2, 4 and 6 in MEG-3 3223, O3020DS nTG, O1035DS nTG and placebo adjusted for intake level.
Additional 2: Change from baseline in plasma phospholipid DHA at weeks 2, 4 and 6 across the treatment groups adjusted for intake level. | Baseline, week 2, week 4, week 6
  Change from baseline in plasma phospholipid DHA at weeks 2, 4 and 6 in MEG-3 3223, O3020DS nTG, O1035DS nTG and placebo adjusted for intake level.
Additional 3: Cytokines/Inflammatory markers | Baseline, week 6
  Exploratory parameters [e.g., Cytokines and inflammatory markers (e.g., TNF-alpha, IL-1alpha, IL1beta, IL-6, IL-10, hs-CRP, HbA1c) will be assessed at baseline and week 6.
Additional 3: Neurotransmitters | Baseline, week 6
  Exploratory parameters: neurotransmitters (e.g., GABA, BDNF, serotonin, cortisol) will be assessed at baseline and week 6.,
Additional 3: Oxylipins | Baseline, week 6
  Exploratory parameters: oxylipins (e.g. resolvins, maresins, protectins) will be assessed at baseline and week 6.
Additional 3: PhenoAgeAccel index | Baseline, week 6
  Exploratory parameters (PhenoAge Accel Index) at baseline and week 6. This is a metric calculated from phenotypic and chronological age, albumin, creatinine, alkaline phosphatase, glycated haemoglobin, WBC count, lymphocyte percentage, haemoglobin, red cell distribution width, MCV and, glucose).
Additional 3: Aging Clock (iAge) | Baseline, week 6
  Exploratory parameters (Aging Clock) at baseline and week 6. This is a metric calculated from CXCL9, CCL11, CCL3, leptin, IL-1beta, IL-5, IFN-alpha, IFN-gamma, IL-4.
Additional 3: PhenoAge Clock | Baseline, week 6
  Exploratory parameters (PhenoAge Clock) at baseline and week 6. An epigenetic clock comprised of DNA methylation (DNAm) algorithms that combine information from measurements across the genome to quantify variations in biological versus chronological aging.
Additional 3: Brain Health Score | Baseline, week 6
  Exploratory parameters (Brain Health Score) at baseline and week 6. Brain health score derived from plasma proteomic and metabolomic biomarkers.
Safety Endpoint 1: Clinical Chemistry | Screening, week 6
  Screening and final visit clinical chemistry profiles will be assessed from a blood sample by a clinical analyser. Tests included in the clinical chemistry profile include sodium, potassium, chloride, bicarbonate, anion gap, calcium (corrected), phosphate, urea, urate, creatinine, eGFR, glucose, total protein, albumin, globulins, total bilirubin, direct bilirubin, alkaline phosphatase (ALP), aspartate transaminase (AST), alanine transaminase (ALT), GGT, lactate dehydrogenase, iron studies, creatine kinase, magnesium, cholesterol, triglycerides, HDL and LDL.
Safety Endpoint 1: Haematology | Screening, week 6
  Screening and final visit haematology profiles will be assessed from a blood sample by a clinical analyser. Tests included in the haematology profile are haemoglobin, MCV, RCC, haematocrit, MCH, MCHC, RDW%, reticulocytes, ESR, platelets, white cell count, neutrophils, lymphocytes, monocytes, eosinophils and basophils.
Safety Endpoint 2: BP | Screening, baseline and week 6
  Vital signs: Blood pressure (BP) will be assessed at screening/baseline and final visit.
Safety Endpoint 2: HR | Screening, baseline, week 6
  Vital signs: Heart rate (HR) will be assessed at screening/baseline and final visit.
Safety Endpoint 2: Body temperature | Screening, baseline, week 6
  Vital signs: Body temperature will be assessed at screening/baseline and final visit.
Safety Endpoint 3: Weight | Screening, baseline, week 6
  Anthropometric: Weight (kg) will be assessed at screening, baseline and the final visit.
Safety Endpoint 3: WHR | Baseline, week 6
  Anthropometric: Waist-hip-ratio (WHR) will be assessed at baseline and the final visit.
Safety Endpoint 4: AEs | Screening to week 6
  Adverse event (AE) listing will be collected.
Safety Endpoint 5: SAEs | Baseline to week 6
  SAEs will be collected and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Birkett, Study Director — dsm-firmenich Switzerland AG
Locations (1):
- RDC Clinical, Fortitude Valley, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study also registered on ISRCTN registry — https://www.isrctn.com/ISRCTN12166286